CLINICAL TRIAL: NCT03691025
Title: Ultrasonographic Measurement of the Optic Nerve Sheath Diameter and Its Association With Eyeball Transverse Diameter in Robot-assisted Laparoscopic Radical Prostatectomy
Brief Title: Association of the Optic Nerve Sheath Diameter With Eyeball Transverse Diameter in Robot-assisted Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Başak Akça, Assist.Prof, Hacettepe University
Other Study IDs: hacetteperobotprostat
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Elevated Intracranial Pressure; Optic Nerve Sheath Diameter; ONSD /ETD Ratio
Keywords: robot assisted laparoscopic prostatectomy; optic nerve sheath diameter
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RALPD

SUMMARY:
Robot-assisted laparoscopic radical prostatectomy (RALRP) is becoming a popular procedure due to its unique advantages.

Despite these advantages, pneumoperitoneum and steep trendelenburg position are associated with hemodynamic instability and elevated intracranial pressures (ICP).

Ultrasonographic measurement of optic nerve sheath diameter (ONSD) is an indirect but also a generally accepted reliable and noninvasive measurement of elevated ICP. However, optimal cut-off values are highly inconsistent due to multiple factors (gender, height, weight). To eliminate the effects of these factors on the results; a ratio should be established in patients known to have elevated ICPs.

In a recent study ONSD/ eyeball transverse diameter(ETD) in healthy volunteers in a specific population was established.

60 patients without any history of ICP undergoing RALRP will be enrolled to the study. Ultrasonographic measurement of ONSD and ETD will be performed 10 minutes after induction of general anesthesia, 10 minutes after CO2 pneumoperitoneum with trendelenburg positioning and measurements will be repeated hourly and at last after returning to supine position without CO2 pneumoperitoneum at the end of the procedure.

Hemodynamic variables and BIS values on this specific times will be recorded and an arterial sample will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* 19-75 years patients undergoing RALP

Exclusion Criteria:

* a history of corneal surgery, open-angle or closed-angle glaucoma
* intraocular surgery
* history of elevated ICPs

Ages: 18 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: patients referred to Hacettepe University Department of Urology
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-02-15 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Association of the Optic Nerve Sheath Diameter With Eyeball Transverse Diameter in Robot-assisted Prostatectomy | 6 months
  To determine a cut off value for ratio of ONSD to ETD in a group known to have elevated ICPs

CONTACTS AND LOCATIONS:
Overall Officials: Başak Akça, Principal Investigator — Hacettepe University Department of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim DH, Jun JS, Kim R. Ultrasonographic measurement of the optic nerve sheath diameter and its association with eyeball transverse diameter in 585 healthy volunteers. Sci Rep. 2017 Nov 21;7(1):15906. doi: 10.1038/s41598-017-16173-z. PMID 29162911